CLINICAL TRIAL: NCT05742776
Title: The Relationship Between Ultrasonographic Findings and Sleep Quality in Patients With Carpal Tunnel Syndrome
Brief Title: The Relationship Between Ultrasonographic Findings and Sleep Quality in Carpal Tunnel Syndrome
Status: Recruiting | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Nuran Eyvaz, Principal Investigator, Afyonkarahisar Health Sciences University
Other Study IDs: CTSPUKI23
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Musculoskeletal Diseases; Median Nerve Disease; Carpal Tunnel Syndrome; Ultrasound; Sleep Quality
Keywords: Carpal Tunnel Syndrome; Ultrasonographic evaluation; Pittsburgh Sleep Quality Index
MeSH Terms: conditions — Musculoskeletal Diseases; Median Neuropathy; Carpal Tunnel Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: CTS Patients
  Interventions: Other: Assessment of Sleep Quality
- Control Group: Healthy Individuals
  Interventions: Other: Assessment of Sleep Quality

INTERVENTIONS:
Other: Assessment of Sleep Quality — Assessment of Sleep Quality
  Groups: Patient Group
Other: Assessment of Sleep Quality — Assessment of Sleep Quality
  Groups: Control Group

SUMMARY:
The aim of our study is to determine the relationship between disease severity and sleep quality in CTS patients and to compare the findings with healthy controls.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is the most common form of entrapment neuropathies. Anatomically, the roof of the carpal tunnel consists of carpal bones, it is located under the transverse carpal ligament, and there are 9 tendon packs of the forearm flexors and the median nerve. Clinically, sensory (paresthesia and hypoesthesia), motor deficits and pain occur in the distribution of the median nerve secondary to mechanical compression and local ischemia.

With the increase in the severity of the disease, entrapment neuropathy, whose symptoms are more pronounced at night, negatively affects the daily life of the person. Waking up at night due to paresthesia is one of the diagnostic criteria for carpal tunnel syndrome. However, the mechanism linking CTS with insomnia is unclear.

The aim of our study is to determine the relationship between disease severity and sleep quality in CTS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CTS according to the criteria of the American Academy of Neurology

Exclusion Criteria:

* Patients with radiculopathy, brachial plexopathy, thoracic outlet syndrome and traumatic nerve injury that may affect the median nerve
* History of Carpal tunnel surgery
* Pregnancy
* Malignancy
* Thyroid diseases
* Amyloidosis
* Systemic lupus erythematosus, Rheumatoid arthritis, Systemic sclerosis, Gout, Dermatomyositis, Polymyositis
* Obstructive sleep apnea

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 90 patients with CTS and 30 patients with gonarthrosis as control group, aged between 20-80 years who applied to our clinic will be included in the study.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 2023.02-2023.05
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | 2023.02-2023.05
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is a frequently used questionnaire for CTS that includes 2 components. It evaluates for grading under two sub-headings: symptom severity scale (11 questions) and functional status scale (8 questions). Scores range from 0 to 5 for each question; 0 represents no difficulty during the activity, 5 represents extremely severe dysfunction.
Cross-sectional area of the Median Nerve (CSA) | 2023.02-2023.05
  The cross-sectional area (CSA) of the median nerve will be used for analysis by the mean value of 3 measurements made with an electronic caliper at scaphoid-pisiform level. Ultrasonographic evaluations were planned to be performed with the 10-18-MHz linear probe of the MyLab 70 (Esaote, Genova, Italy) device by a physician experienced in US.
  CSA values increase as clinical findings worsen.
Electrophysiological Evaluation | 2023.02-2023.05
  The patients will be evaluated as mild-moderate-severe CTS according to the criteria of the American Academy of Neurology.
Hand and Finger Grip Strength Assessment | 2023.02-2023.05
  The hand grip strength of the participants will be measured with the "Jamar Hand Dynamometer". Measurements will be made with the shoulder in adduction and neutral rotation adjacent to the trunk, elbow 90 degrees flexed, wrist 0-30 degrees dorsiflexion and 0-15 degrees ulnar deviation with thumb up. Finger grip strength will be evaluated with the "Jamar Digital Pinchmeter". Patients will be placed in the sitting position with the wrist in 90° flexion and the forearm in the neutral position. Measurements will be made bilaterally in three different positions as lateral, palmar and fingertip grips. Patients will be asked to squeeze with maximum force and each measurement will be made three times, and their averages will be recorded in kg. The dynamometer has a dual scale readout which displays isometric grip force from 0-90 kg. Higher scores means better grip strength.
Pittsburgh Sleep Quality Index (PSQI) | 2023.02-2023.05
  Pittsburgh Sleep Quality Index (PSQI) is a questionnaire that assesses sleep patterns and sleep quality in adults. The measure consists subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping pills, and daytime dysfunction in the past month. The global score of PUKI and each sub-parameter will be calculated and recorded separately. According to the PSQI, "good sleepers" are defined as a PSQI score = <5 and "bad sleepers" as PSQI > 5.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University; Ali İzzet AKÇİN, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Afyonkarahi̇sar, Turkey (Türkiye)

REFERENCES:
- [Background] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Background] Okkesim CE, Serbest S, Tiftikci U, Cirpar M. Prospective evaluation of preoperative and postoperative sleep quality in carpal tunnel release. J Hand Surg Eur Vol. 2019 Mar;44(3):278-282. doi: 10.1177/1753193418808182. Epub 2018 Nov 4. PMID 30394830
- [Background] Kaymak B, Ozcakar L, Cetin A, Candan Cetin M, Akinci A, Hascelik Z. A comparison of the benefits of sonography and electrophysiologic measurements as predictors of symptom severity and functional status in patients with carpal tunnel syndrome. Arch Phys Med Rehabil. 2008 Apr;89(4):743-8. doi: 10.1016/j.apmr.2007.09.041. PMID 18374007